CLINICAL TRIAL: NCT04447287
Title: Phase 1b Randomized, Placebo-controlled Study to Assess the Effect of a Single Dose of ASP8062 on the Multiple Dose Safety, Tolerability and Pharmacokinetics of Buprenorphine/Naloxone in Subjects With Opioid Use Disorder
Brief Title: A Study to Assess the Effect of a Single Dose of ASP8062 on the Multiple Dose Safety, Tolerability and Pharmacokinetics of Buprenorphine/Naloxone in Participants With Opioid Use Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8062-CL-2003; UG3DA051392 (NIH)
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Results first posted 2022-01-12 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Opioid Use Disorder
Keywords: Suboxone®; Opioid Use Disorder; buprenorphine/naloxone; ASP8062; pharmacokinetic
MeSH Terms: conditions — Opioid-Related Disorders | interventions — ASP8062; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ASP8062 in combination with buprenorphine/naloxone (Experimental): Participants received multiple sublingual doses of buprenorphine/naloxone on days 1 through 26. In the Investigational Period participants were on a stable daily dose of buprenorphine/naloxone on days 5 through 18. After randomization on day 12, participants received a single oral dose of ASP8062 concomitantly with buprenorphine/naloxone. The stable dose of buprenorphine/naloxone was down titrated from days 19 through 26.
  Interventions: Drug: ASP8062; Drug: buprenorphine/naloxone
- Placebo ASP8062 in combination with buprenorphine/naloxone (Placebo Comparator): Participants received multiple sublingual doses of buprenorphine/naloxone on days 1 through 26. In the Investigational Period participants were on a stable daily dose of buprenorphine/naloxone on days 5 through 18. After randomization on day 12, participants received a single oral dose of placebo concomitantly with buprenorphine/naloxone. The stable dose of buprenorphine/naloxone was down titrated from days 19 through 26.
  Interventions: Drug: Placebo ASP8062; Drug: buprenorphine/naloxone

INTERVENTIONS:
Drug: ASP8062 — Oral
  Arms: ASP8062 in combination with buprenorphine/naloxone
Drug: Placebo ASP8062 — Oral
  Arms: Placebo ASP8062 in combination with buprenorphine/naloxone
Drug: buprenorphine/naloxone — Sublingual
  Other Names: Suboxone®

SUMMARY:
The primary purpose of this study was to assess the safety and tolerability of multiple doses of buprenorphine/naloxone alone and buprenorphine/naloxone in combination with a single dose of ASP8062.

This study also assessed the potential for pharmacokinetic interaction between ASP8062 and buprenorphine/naloxone.

DETAILED DESCRIPTION:
Participants were screened for up to 28 days prior to first investigational product (IP) administration. Eligible participants were admitted to the clinical unit on day -1 and were residential for a single period of 27 days/26 nights.

Participants were discharged from the clinical unit after completion of down-titration on the condition that all required assessments were performed and that there were no medical reasons for a longer stay in the clinical unit; which was the end-of-study visit (ESV). Prior to discharge, participants were provided with local buprenorphine and methadone providers for their reference.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index range of 18 to 36 kg/m^2, inclusive and weighs at least 50 kg at screening.
* Subject has a diagnosis of moderate or severe opioid use disorder (OUD) according to the Diagnostic and Statistical Manual of Mental Disorders, edition 5 (DSM-5) at screening.
* Subject tests positive for opioids at screening and/or on day -1 or subject shows signs of opioid withdrawal on day -1.
* Subject is willing to take buprenorphine/naloxone and is not taking buprenorphine or buprenorphine/naloxone at screening.
* Female subject is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 30 days after final investigational product (IP) administration.
* Female subject must agree not to breastfeed starting at screening and throughout the study period and for 30 days after final IP administration.
* Female subject must not donate ova starting at first dose of IP and throughout the study period and for 30 days after final IP administration.
* Male subject with female partner(s) of childbearing potential (including breastfeeding partner) must agree to use contraception throughout the study period and for 90 days after final IP administration.
* Male subject must not donate sperm during the treatment period and for 90 days after final IP administration.
* Male subject with pregnant partner(s) must agree to remain abstinent or use a condom and spermicide for the duration of the pregnancy throughout the study period and for 90 days after final IP administration.
* Subject agrees not to participate in another interventional study while participating in the present study.
* Subject must be willing to abstain from smoking (including use of tobacco containing products and nicotine or nicotine-containing products [e.g., electronic vapes] from at least 1 hour predose through at least 8 hours postdose on days 11 and 12.

Exclusion Criteria:

* Subject has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Subject has any condition which makes the subject unsuitable for study participation.
* Female subject who has been pregnant within 6 months prior to screening or breastfeeding within 3 months prior to screening.
* Subject has a known or suspected hypersensitivity to ASP8062, buprenorphine, naloxone or any components of the formulations used.
* Subject has had previous exposure with ASP8062.
* Subject has any of the liver function tests (alkaline phosphatase [ALP], alanine aminotransferase [ALT], aspartate aminotransferase [AST], gamma-glutamyl transferase and total bilirubin [TBL]) > 2 × upper limit of normal (ULN) on day -1. In such a case, the assessment may be repeated once.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies) prior to first IP administration.
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, renal and/or other major disease or malignancy with exception of history of cholecystectomy.
* Subject has current or recent diagnosis (within the last 12 months) of moderate or severe alcohol, sedative, hypnotic, anxiolytic, cocaine or any other substance use disorder (except for opioids, caffeine, tobacco or nicotine) according to the DSM-5 at screening.
* Subject has a history or presence of any clinically significant psychiatric disorders such as, bipolar 1, schizophrenia, schizoaffective disorder or major depressive disorders.
* Subject tests positive for alcohol, benzodiazepine or methadone on day -1. Subject tests positive for buprenorphine on day -1.
* Subject has had recent suicidal ideation within the last 12 months or subject who is at significant risk to commit suicide using the Columbia-Suicide Severity Rating Scale (C-SSRS) at screening or since the last visit on day -1.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 1 week prior to day -1.
* Subject has any clinically significant abnormality following physical examination, electrocardiogram (ECG) and protocol-defined clinical laboratory tests at screening or on day -1.
* Subject has a mean pulse < 45 or > 110 beats per minute (unless out of range [> 110 beats per minute] pulse is deemed to be secondary to opioid withdrawal); mean systolic blood pressure > 150 mmHg; mean diastolic blood pressure > 95 mmHg (unless out of range blood pressure is deemed to be secondary to opioid withdrawal)(measurements taken in duplicate after subject has been resting in the supine position for at least 5 minutes; pulse will be measured automatically) on day -1. If the mean blood pressure exceeds the limits above, 1 additional duplicate may be taken.
* Subject has a mean corrected QT interval using Fridericia's formula (QTcF) of > 450 msec (for male subjects) and > 470 msec (for female subjects) on day -1. If the mean QTcF exceeds the limits above, 1 additional duplicate ECG may be taken.
* Subject has used any prescribed drugs, vitamins and natural or herbal remedies (including, St. John's Wort) in the 2 weeks prior to first IP administration, except for rescue medications, milk of magnesia, acetaminophen, topical dermatological products, including corticosteroid products, hormonal contraceptives and hormone replacement therapy (HRT).
* Subject has used any inducer of metabolism (e.g., barbiturates and rifampin) in the 3 months prior to day -1.
* Subject has had significant blood loss or donated approximately 500 mL of whole blood (excluding plasma donation) within 56 days prior to screening or donated plasma within 7 days prior to day -1.
* Subject has a positive serology test for antibodies to human immunodeficiency virus type 1 and/or type 2, acute hepatitis B virus infection or acute hepatitis C virus infection, excluding asymptomatic hepatitis C virus infection at screening.
* Subject has loss of ability to freely provide consent through imprisonment or involuntary incarceration for treatment of either a psychiatric or physical (e.g., infectious disease) illness.
* Subject is an employee of Astellas, the study-related contract research organizations or the clinical unit.
* Subject has used any inducer of CYP2C8, 2C9 or 3A4-related metabolism (e.g., barbiturates, rifampin, aprepitant, ritonavir, apalutamide, carbamazepine, enzalutamide, mitotane, phenytoin, rifampin, St. John's wort, bosentan, efavirenz, etravirine, phenobarbital, primidone, armodafinil, modafinil, and rufinamide) in the 3 months prior to day -1.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Altasciences Clinical Kansas, Inc., Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Ito M, Walzer M, Beth Blauwet M, Spence A, Heo N, Kelsh D, Blahunka P, Erdman J, Nour Alsharif M, Marek GJ. A phase 1b study to investigate the potential interactions between ASP8062 and buprenorphine/naloxone in patients with opioid use disorder. J Psychopharmacol. 2023 Feb;37(2):144-154. doi: 10.1177/02698811221149657. Epub 2023 Feb 3. PMID 36738100
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/8062-CL-2003/
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14687&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who had opioid use disorder (OUD) were enrolled in this study. Participants were enrolled in one site in the United States.
Pre-assignment Details: Participants were randomized using a 2:1 ratio. Eligible participants who met inclusion criteria and none of the exclusion criteria were enrolled. A total of 74 participants entered the screening process and out of which 56 discontinued prior to randomization. Prior to randomization, participants entered a run-in period. A total of 23 participants entered the run-in period and 19 completed, 1 participant completed the run-in period but discontinued before randomization.
Groups:
- Buprenorphine/Naloxone: Participants received multiple sublingual doses of buprenorphine/naloxone on days 1 through 26. Participants were on a stable daily dose of buprenorphine/naloxone on days 5 through 18. The stable dose of buprenorphine/naloxone was down titrated from days 19 through 26.
Period: Period 1: Run-in Period
Arm/Group | Buprenorphine/Naloxone | ASP8062 in Combination With Buprenorphine/Naloxone | Placebo ASP8062 in Combination With Buprenorphine/Naloxone
Started | 23 | 0 | 0
Completed | 19 | 0 | 0
Not Completed | 4 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Period 2: Investigational Period
Arm/Group | Buprenorphine/Naloxone | ASP8062 in Combination With Buprenorphine/Naloxone | Placebo ASP8062 in Combination With Buprenorphine/Naloxone
Started | 1 | 12 | 6
Completed | 0 | 12 | 6
Not Completed | 1 | 0 | 0
Not completed — Completed the run-in period but discontinued before randomization due to limited samples collected. | 1 | 0 | 0
Period: Period 3: Down-Titration Period
Arm/Group | Buprenorphine/Naloxone | ASP8062 in Combination With Buprenorphine/Naloxone | Placebo ASP8062 in Combination With Buprenorphine/Naloxone
Started | 0 | 12 | 6
Completed | 0 | 12 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population consisted of all participants who received at least 1 dose of Investigational Product (IP) during Run-in Period; Investigational Period and Down-titration Period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Buprenorphine/Naloxone | ASP8062 in Combination With Buprenorphine/Naloxone | Placebo ASP8062 in Combination With Buprenorphine/Naloxone | Total
Number analyzed (Participants) | 5 | 12 | 6 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.4 (5.2) | 40.2 (9.2) | 43.2 (10.3) | 41.2 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 7
  Male | 3 | 9 | 4 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 12 | 6 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 7 | 5 | 16
  White | 1 | 5 | 1 | 7
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Blood Oxygen Saturation (SpO2) [Mean (Standard Deviation); unit: percentage of oxygen saturation] — The SpO2 was measured using a pulse oximeter placed on the participant's fingertip. Baseline for SpO2 measurement was the last non-missing observation prior to first administration of Investigational Product (IP). Population: The analysis population consisted of all participants who received at least 1 dose of IP during Run-in Period; Investigational Period and Down-titration Period.
  percentage of oxygen saturation
    number analyzed (Participants) | 5 | 11 | 6 | 22
    (all) | 98.2 (0.8) | 97.8 (1.9) | 97.8 (1.2) | 97.9 (1.5)
End Tidal Carbon Dioxide (CO2) [Mean (Standard Deviation); unit: millimeter of mercury (mmHg)] — End tidal CO2 measurement was obtained per participant utilizing a portable bedside capnography device. The baseline is study Day 11, prior to dosing with ASP8062 or Placebo ASP8062. Population: The analysis population consisted of all participants who received at least 1 dose of IP during Run-in Period; Investigational Period and Down-titration Period.
  millimeter of mercury (mmHg)
    number analyzed (Participants) | 1 | 12 | 6 | 19
    (all) | 40 (0) | 40.4 (4.1) | 38.2 (5.1) | 39.7 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a participant administered an Investigational Product (IP) and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding; abnormal laboratory test result or other safety assessment, symptom, or disease temporally associated with the use of IP whether or not considered related to the IP. A treatment-emergent adverse event (TEAE) was defined as an AE with onset at any time from first dosing until last scheduled procedure. AEs were considered serious (SAEs) if the AE resulted in death, was life-threatening, resulted in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, resulted in congenital anomaly, or birth defect or required inpatient hospitalization or led to prolongation of hospitalization.
Time Frame: From first dose of study drug up to end of study visit (up to day 27)
Population: The analysis population was the Safety Analysis Set (SAF), which consisted of all participants who received at least 1 dose of ASP8062.
Measure: Number; unit: Participants
Groups:
- Buprenorphine/Naloxone (Run-in Period): Participants received multiple sublingual doses of buprenorphine/naloxone on days 1 through 26. Participants were on a stable daily dose of buprenorphine/naloxone on days 5 through 18. The stable dose of buprenorphine/naloxone was down titrated from days 19 through 26.
- ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period): Participants received multiple sublingual doses of buprenorphine/naloxone on days 12 through 18. After randomization on day 12, participants received a single oral dose of ASP8062 concomitantly with buprenorphine/naloxone and underwent repeat intensive safety assessment on day 12.
- ASP8062 in Combination With Buprenorphine/Naloxone (Down-titration Period): Participants received multiple sublingual doses of buprenorphine/naloxone on days 19 through 26. After randomization on day 12, participants received a single oral dose of ASP8062 concomitantly with buprenorphine/naloxone and underwent repeat intensive safety assessment on day 12. The stable dose of buprenorphine/naloxone was down titrated from days 19 through 26.
- Placebo ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period): Participants received multiple sublingual doses of buprenorphine/naloxone on days 12 through 18. After randomization on day 12, participants received a single oral dose of Placebo concomitantly with buprenorphine/naloxone and underwent repeat intensive safety assessment on day 12.
- Placebo ASP8062 in Combination With Buprenorphine/Naloxone (Down-titration Period): Participants received multiple sublingual doses of buprenorphine/naloxone on days 19 through 26. After randomization on day 12, participants received a single oral dose of Placebo concomitantly with buprenorphine/naloxone and underwent repeat intensive safety assessment on day 12. The stable dose of buprenorphine/naloxone was down titrated from days 19 through 26.
Arm/Group | Buprenorphine/Naloxone (Run-in Period) | ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period) | ASP8062 in Combination With Buprenorphine/Naloxone (Down-titration Period) | Placebo ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period) | Placebo ASP8062 in Combination With Buprenorphine/Naloxone (Down-titration Period)
Number analyzed (Participants) | 23 | 12 | 12 | 6 | 6
Participants
  TEAE | 16 | 6 | 7 | 6 | 2
  Drug-Related TEAE | 12 | 6 | 5 | 6 | 1
  Serious TEAE | 0 | 0 | 0 | 0 | 0
  Drug-Related Serious TEAE | 0 | 0 | 0 | 0 | 0
  TEAE Leading to Death | 0 | 0 | 0 | 0 | 0
  Drug-Related TEAE Leading to Death | 0 | 0 | 0 | 0 | 0
  TEAE Leading to Withdrawal of Treatment | 0 | 0 | 0 | 0 | 0
  Drug-Related TEAE Leading to Withdrawal of Treatment | 0 | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Suicidal Ideation and/or Suicidal Behavior as Assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS) is a clinician administered assessment tool that evaluates suicidal ideation and behavior. Number of participants that have an affirmative response to the 5 items for suicidal ideation (1. Wish to be dead, 2. Non-specific active suicidal thoughts, 3. Active suicidal ideation with any methods (not plan) without intent to act, 4. Active suicidal ideation with some intent to act, without specific plan, 5. Active suicidal ideation with specific plan and intent) and/or to the 5 items for suicidal behavior (1. Preparatory acts or behavior, 2. Aborted attempt, 3. Interrupted attempt, 4. Actual attempt, 5. Completed suicide) were reported.
Time Frame: Up to day 27
Population: The analysis population was the SAF, which consisted of all participants who received at least 1 dose of Investigational Product (IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Buprenorphine/Naloxone (Run-in Period) | ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period) | ASP8062 in Combination With Buprenorphine/Naloxone (Down-titration Period) | Placebo ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period) | Placebo ASP8062 in Combination With Buprenorphine/Naloxone (Down-titration Period)
Number analyzed (Participants) | 23 | 12 | 12 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Change From Baseline in Blood Oxygen Saturation (SpO2) at Predose
Description: The blood oxygen saturation (SpO2 was measured using a pulse oximeter placed on the participant's fingertip. Change from baseline in SpO2 was calculated as Day 11 minus Baseline for arm 'buprenorphine/naloxone', and Day 12 minus Baseline for arms 'ASP8062 in combination with buprenorphine/naloxone' and 'Placebo ASP8062 in combination with buprenorphine/naloxone'. Baseline observation was last non-missing observation prior to first dose.
Time Frame: 'buprenorphine/naloxone': Baseline and 1 hour postdose Day 11; 'ASP8062 in combination with buprenorphine/naloxone' and 'Placebo ASP8062 in combination with buprenorphine/naloxone': Baseline and 1 hour postdose Day 12
Population: The analysis population was the SAF, which consisted of all participants who received at least 1 dose of IP and had baseline and post dose measures taken. It was pre-specified to assess only the Run-in Period and Investigational Period Arms/Groups for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: Percentage of oxygen saturation
Arm/Group | Buprenorphine/Naloxone (Run-in Period) | ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period) | Placebo ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period)
Number analyzed (Participants) | 18 | 11 | 6
Percentage of oxygen saturation | 0.2 (2.1) | -0.4 (2.3) | -0.3 (1.9)

4. Primary Outcome: Change From Baseline in Blood Oxygen Saturation (SpO2) at 1 Hour Postdose
Description: The blood oxygen saturation (SpO2) was measured using a pulse oximeter placed on the participant's fingertip. Change from baseline in SpO2 was calculated as Day 11 minus Baseline for arm 'buprenorphine/naloxone', and Day 12 minus Baseline for arms 'ASP8062 in combination with buprenorphine/naloxone' and 'Placebo ASP8062 in combination with buprenorphine/naloxone'. Baseline observation was last non-missing observation prior to first dose.
Time Frame: as for outcome 3
Population: The analysis population was the SAF, which consisted of all participants who received at least 1 dose of IP and had both baseline and post dose measures taken. It was pre-specified to assess only the Run-in Period and Investigational Period Arms/Groups for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: Percentage of oxygen saturation
Arm/Group | Buprenorphine/Naloxone (Run-in Period) | ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period) | Placebo ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period)
Number analyzed (Participants) | 18 | 11 | 6
Percentage of oxygen saturation | 0.1 (2.5) | -0.6 (2.6) | -0.7 (2.3)

5. Primary Outcome: Change From Baseline in Blood Oxygen Saturation (SpO2) at 2 Hour Postdose
Description: as for outcome 4
Time Frame: 'buprenorphine/naloxone': Baseline and 2 hour postdose Day 11; 'ASP8062 in combination with buprenorphine/naloxone' and 'Placebo ASP8062 in combination with buprenorphine/naloxone': Baseline and 2 hour postdose Day 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of oxygen saturation
Arm/Group | Buprenorphine/Naloxone (Run-in Period) | ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period) | Placebo ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period)
Number analyzed (Participants) | 18 | 11 | 6
Percentage of oxygen saturation | 0.2 (2.2) | -0.8 (2.0) | 0.3 (1.8)

6. Primary Outcome: Change From Baseline in Blood Oxygen Saturation (SpO2) at 4 Hour Postdose
Description: as for outcome 4
Time Frame: 'buprenorphine/naloxone': Baseline and 4 hour postdose Day 11; 'ASP8062 in combination with buprenorphine/naloxone' and 'Placebo ASP8062 in combination with buprenorphine/naloxone': Baseline and 4 hour postdose Day 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of oxygen saturation
Arm/Group | Buprenorphine/Naloxone (Run-in Period) | ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period) | Placebo ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period)
Number analyzed (Participants) | 18 | 11 | 6
Percentage of oxygen saturation | 0.3 (1.9) | -0.4 (1.7) | -0.2 (1.2)

7. Primary Outcome: Change From Baseline in Blood Oxygen Saturation (SpO2) at 8 Hour Postdose
Description: as for outcome 4
Time Frame: 'buprenorphine/naloxone': Baseline and 8 hour postdose Day 11; 'ASP8062 in combination with buprenorphine/naloxone' and 'Placebo ASP8062 in combination with buprenorphine/naloxone': Baseline and 8 hour postdose Day 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of oxygen saturation
Arm/Group | Buprenorphine/Naloxone (Run-in Period) | ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period) | Placebo ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period)
Number analyzed (Participants) | 18 | 11 | 6
Percentage of oxygen saturation | 0.1 (2.3) | -0.1 (2.4) | 0.7 (1.6)

8. Primary Outcome: Change From Baseline in Blood Oxygen Saturation (SpO2) at 12 Hour Postdose
Description: as for outcome 4
Time Frame: 'buprenorphine/naloxone': Baseline and 12 hour postdose Day 11; 'ASP8062 in combination with buprenorphine/naloxone' and 'Placebo ASP8062 in combination with buprenorphine/naloxone': Baseline and 12 hour postdose Day 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of oxygen saturation
Arm/Group | Buprenorphine/Naloxone (Run-in Period) | ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period) | Placebo ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period)
Number analyzed (Participants) | 18 | 11 | 6
Percentage of oxygen saturation | -0.6 (1.8) | -0.3 (2.5) | -0.5 (0.8)

9. Primary Outcome: Change From Baseline in End Tidal Carbon Dioxide (CO2) at Predose
Description: End tidal CO2 measurements was obtained per participant utilizing a portable bedside capnography device. Change from baseline in CO2 was calculated as Day 12 minus Baseline for arms 'ASP8062 in combination with buprenorphine/naloxone' and 'Placebo ASP8062 in combination with buprenorphine/naloxone'.
Time Frame: 'ASP8062 in combination with buprenorphine/naloxone' and 'Placebo ASP8062 in combination with buprenorphine/naloxone': Baseline and predose Day 12
Population: The analysis population was the Safety Analysis Set (SAF), which consisted of all participants who received at least 1 dose of ASP8062. It was pre-specified to assess only the Investigational Period Arms/Groups for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period) | Placebo ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period)
Number analyzed (Participants) | 12 | 6
mmHg | -1.3 (4.0) | 0.5 (6.1)

10. Primary Outcome: Change From Baseline in End Tidal Carbon Dioxide (CO2) at 1 Hour Postdose
Description: End tidal CO2 measurements was obtained per participant utilizing a portable bedside capnography device. Change from baseline in CO2 was calculated as Day 11 minus Baseline for arm 'buprenorphine/naloxone', and Day 12 minus Baseline for arms 'ASP8062 in combination with buprenorphine/naloxone' and 'Placebo ASP8062 in combination with buprenorphine/naloxone'.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Buprenorphine/Naloxone (Run-in Period) | ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period) | Placebo ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period)
Number analyzed (Participants) | 19 | 12 | 6
mmHg | 1.3 (5.8) | -0.5 (4.0) | 3.7 (7.2)

11. Primary Outcome: Change From Baseline in End Tidal Carbon Dioxide (CO2) at 2 Hour Postdose
Description: as for outcome 10
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Buprenorphine/Naloxone (Run-in Period) | ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period) | Placebo ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period)
Number analyzed (Participants) | 19 | 12 | 6
mmHg | 1.2 (5.1) | 0.3 (3.2) | 4.2 (5.0)

12. Primary Outcome: Change From Baseline in End Tidal Carbon Dioxide (CO2) at 4 Hour Postdose
Description: as for outcome 10
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Buprenorphine/Naloxone (Run-in Period) | ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period) | Placebo ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period)
Number analyzed (Participants) | 18 | 12 | 6
mmHg | 0.9 (4.9) | -1.0 (2.3) | 5.3 (7.9)

13. Primary Outcome: Change From Baseline in End Tidal Carbon Dioxide (CO2) at 8 Hour Postdose
Description: as for outcome 10
Time Frame: as for outcome 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Buprenorphine/Naloxone (Run-in Period) | ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period) | Placebo ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period)
Number analyzed (Participants) | 18 | 12 | 6
mmHg | 3.1 (4.1) | 1.4 (1.9) | 6.0 (5.7)

14. Secondary Outcome: Pharmacokinetics (PK) of ASP8062 in Plasma: Area Under the Concentration-time Curve From the Time of Dosing Extrapolated to Time Infinity (AUCinf)
Description: AUCinf was recorded from the PK plasma samples collected. Samples for AUCinf were collected for arm 'ASP8062 in combination with buprenorphine/naloxone' at Day 12.
Time Frame: Predose on day 12 and at the following postdose time points on day 12: 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120, 144, 168, 216 and 264 hour(s)
Population: The analysis population was the Pharmacokinetic Analysis Set (PKAS), which consisted of all participants who received at least 1 dose of ASP8062 for which concentration data was available to facilitate derivation of at least 1 primary pharmacokinetic parameter.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | ASP8062 in Combination With Buprenorphine/Naloxone
Number analyzed (Participants) | 12
h*ng/mL | 4450 (1750)

15. Secondary Outcome: Pharmacokinetics (PK) of ASP8062 in Plasma: Area Under the Concentration-time Curve From the Time of Dosing to the Last Measurable Concentration (AUClast)
Description: AUClast was recorded from the PK plasma samples collected. Samples for AUClast were collected for arm 'ASP8062 in combination with buprenorphine/naloxone' at Day 12.
Time Frame: as for outcome 14
Population: The analysis population was the PKAS, which consisted of all participants who received at least 1 dose of ASP8062 for which concentration data was available to facilitate derivation of at least 1 primary pharmacokinetic parameter.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | ASP8062 in Combination With Buprenorphine/Naloxone
Number analyzed (Participants) | 12
h*ng/mL | 4270 (1620)

16. Secondary Outcome: Pharmacokinetics (PK) of ASP8062 in Plasma: Maximum Concentration (Cmax)
Description: Cmax was recorded from the PK plasma samples collected. Samples for Cmax were collected for arm 'ASP8062 in combination with buprenorphine/naloxone' at Day 12.
Time Frame: as for outcome 14
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ASP8062 in Combination With Buprenorphine/Naloxone
Number analyzed (Participants) | 12
ng/mL | 152 (36.7)

17. Secondary Outcome: Pharmacokinetics (PK) of Buprenorphine in Plasma: Area Under the Concentration-time Curve From the Time of Dosing to 24 Hours (AUC24)
Description: AUC24 was recorded from the PK plasma samples collected. Samples for AUC24 were collected for arm 'buprenorphine/naloxone' at Day 11; 'ASP8062 in combination with buprenorphine/naloxone' and 'ASP8062 in combination with Placebo' at Day 12.
Time Frame: Predose on day 11 and at the following postdose time points on day 11: 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12 and 16 hour(s)
Population: The analysis population was the PKAS, which consisted of all participants who received at least 1 dose of buprenorphine (in any applicable period) and for which concentration data were available to facilitate derivation of at least 1 primary pharmacokinetic parameter.
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | Buprenorphine/Naloxone | ASP8062 in Combination With Buprenorphine/Naloxone | Placebo ASP8062 in Combination With Buprenorphine/Naloxone
Number analyzed (Participants) | 15 | 12 | 6
h*pg/mL | 63800 (20300) | 53500 (18300) | 67700 (18700)
Statistical Analysis 1: Comparison: Buprenorphine/Naloxone vs ASP8062 in Combination With Buprenorphine/Naloxone; Test type: Other; Geometric LS Mean Ratio = 89.72, 90% CI 2-sided [81.21 to 99.11]

18. Secondary Outcome: Pharmacokinetics (PK) of Buprenorphine in Plasma: Cmax
Description: Cmax was recorded from the PK plasma samples collected. Samples for Cmax were collected for arm 'buprenorphine/naloxone' at Day 11; 'ASP8062 in combination with buprenorphine/naloxone' and 'ASP8062 in combination with Placebo' at Day 12.
Time Frame: Predose on day 11 and at the following postdose time points on day 11: 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12 and 16 hour(s)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Buprenorphine/Naloxone | ASP8062 in Combination With Buprenorphine/Naloxone | Placebo ASP8062 in Combination With Buprenorphine/Naloxone
Number analyzed (Participants) | 18 | 12 | 6
pg/mL | 7790 (3280) | 6790 (3230) | 8440 (2200)
Statistical Analysis 1: Comparison: Buprenorphine/Naloxone vs ASP8062 in Combination With Buprenorphine/Naloxone; Test type: Other; Geometric LS Mean Ratio = 92.15, 90% CI 2-sided [80.22 to 105.86]

19. Secondary Outcome: Pharmacokinetics (PK) of Norbuprenorphine (Buprenorphine's Metabolite) in Plasma: AUC24
Description: as for outcome 17
Time Frame: Predose on day 11 and at the following postdose time points on day 11: 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12 and 16 hour(s)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | Buprenorphine/Naloxone | ASP8062 in Combination With Buprenorphine/Naloxone | Placebo ASP8062 in Combination With Buprenorphine/Naloxone
Number analyzed (Participants) | 15 | 12 | 6
h*pg/mL | 97600 (49200) | 96200 (45700) | 104000 (43600)
Statistical Analysis 1: Comparison: Buprenorphine/Naloxone vs ASP8062 in Combination With Buprenorphine/Naloxone; Test type: Other; Geometric LS Mean Ratio = 109.09, 90% CI 2-sided [101.10 to 117.71]

20. Secondary Outcome: Pharmacokinetics (PK) of Norbuprenorphine (Buprenorphine's Metabolite) in Plasma: Cmax
Description: as for outcome 18
Time Frame: Predose on day 11 and at the following postdose time points on day 11: 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12 and 16 hour(s)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Buprenorphine/Naloxone | ASP8062 in Combination With Buprenorphine/Naloxone | Placebo ASP8062 in Combination With Buprenorphine/Naloxone
Number analyzed (Participants) | 18 | 12 | 6
pg/mL | 5260 (2350) | 6060 (2870) | 5730 (1930)
Statistical Analysis 1: Comparison: Buprenorphine/Naloxone vs ASP8062 in Combination With Buprenorphine/Naloxone; Test type: Other; Geometric LS Mean Ratio = 117.77, 90% CI 2-sided [106.41 to 130.34]

21. Secondary Outcome: Pharmacokinetics (PK) of Naloxone in Plasma: AUC24
Description: as for outcome 17
Time Frame: Predose on day 12 and at the following postdose time points on day 12: 0.25, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 16, 24, 168, 216 and 264 hour(s)
Population: The analysis population was the PKAS, which consisted of all participants who received at least 1 dose of naloxone (in any applicable period) and for which concentration data were available to facilitate derivation of at least 1 primary pharmacokinetic parameter.
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | Buprenorphine/Naloxone | ASP8062 in Combination With Buprenorphine/Naloxone | Placebo ASP8062 in Combination With Buprenorphine/Naloxone
Number analyzed (Participants) | 16 | 12 | 6
h*pg/mL | 1270 (656) | 1060 (624) | 1090 (379)
Statistical Analysis 1: Comparison: Buprenorphine/Naloxone vs ASP8062 in Combination With Buprenorphine/Naloxone; Test type: Other; Geometric LS Mean Ratio = 79.39, 90% CI 2-sided [68.10 to 92.55]

22. Secondary Outcome: Pharmacokinetics (PK) of Naloxone in Plasma: Cmax
Description: as for outcome 18
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Buprenorphine/Naloxone | ASP8062 in Combination With Buprenorphine/Naloxone | Placebo ASP8062 in Combination With Buprenorphine/Naloxone
Number analyzed (Participants) | 18 | 12 | 6
pg/mL | 464 (355) | 382 (284) | 363 (160)
Statistical Analysis 1: Comparison: Buprenorphine/Naloxone vs ASP8062 in Combination With Buprenorphine/Naloxone; Test type: Other; Geometric LS Mean Ratio = 74.45, 90% CI 2-sided [59.28 to 93.50]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to end of study visit (up to day 27)
Arm/Group | Buprenorphine/Naloxone | ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period) | ASP8062 in Combination With Buprenorphine/Naloxone (Down-titration Period) | Placebo ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period) | Placebo ASP8062 in Combination With Buprenorphine/Naloxone (Down-titration Period)
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/12 | 0/12 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/12 | 0/12 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 16/23 | 6/12 | 7/12 | 6/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine/Naloxone (N=23) | ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period) (N=12) | ASP8062 in Combination With Buprenorphine/Naloxone (Down-titration Period) (N=12) | Placebo ASP8062 in Combination With Buprenorphine/Naloxone (Investigational Period) (N=6) | Placebo ASP8062 in Combination With Buprenorphine/Naloxone (Down-titration Period) (N=6)
Constipation (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Feeling of relaxation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 8 (13) | 4 (5) | 2 (3) | 3 (4) | 2 (4)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT04447287/Prot_SAP_000.pdf